CLINICAL TRIAL: NCT00071760
Title: A 48 Week, Phase II, Open-label, 2-cohort, Multicenter Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Antiviral Activity of GW433908 and GW433908/RTV When Administered to HIV-1 Infected Protease Inhibitor (PI) Naive and PI-experienced Pediatric Subjects Aged 4 Weeks to <2 Years.
Brief Title: Study Of An Investigational Regimen Including FDA Approved HIV Drugs In HIV-Infected Pediatric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APV20002
Record Dates: First submitted 2003-10-30; First posted 2003-10-31 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: pediatrics; ritonavir; amprenavir; AGENERASE; HIV; Lexiva; protease inhibitors; HIV Infection; fosamprenavir
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — fosamprenavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - 4weeks - less than 2 years old (FPV/RTV bid) (Experimental): Cohort 2A - 4weeks - less than 6 months old. Fosamprenavir (FPV) 50 mg/mL oral suspension/ritonavir (RTV) 80 mg/mL oral solution twice daily (BID)
  Cohort 1A - 6 months - less than 2yrs old. Fosamprenavir (FPV) 50 mg/mL oral suspension/ritonavir (RTV) 80 mg/mL oral solution twice daily (BID)
  Interventions: Drug: GW433908; Drug: ritonavir
- Arm B- 4weeks - less than 2 years old (FPV bid) (Experimental): Cohort 2B - 4weeks - less than 6 months old. Fosamprenavir (FPV) 50 mg/mL oral suspension twice daily (BID)
  Cohort 1B - 6 months - less than 2yrs old. Fosamprenavir (FPV) 50 mg/mL oral suspension twice daily (BID)
  Interventions: Drug: GW433908

INTERVENTIONS:
Drug: GW433908 — Fosamprenavir suspension bid
Drug: ritonavir — Ritonavir solution bid
  Other Names: GW433908
  Arms: Arm A - 4weeks - less than 2 years old (FPV/RTV bid)

SUMMARY:
This is a 48-week study to evaluate the safety, tolerability, pharmacokinetics, and antiviral activity of an investigational regimen including FDA approved HIV drugs in HIV-infected pediatric subjects, ages 4 weeks to < 2 years old.

DETAILED DESCRIPTION:
A 48 week, Phase II, open-label, 2-cohort, multicenter study to evaluate the pharmacokinetics, safety, tolerability and antiviral activity of GW433908 and GW433908/RTV when administered to HIV-1 infected protease inhibitor (PI) naive and PI-experienced pediatric subjects aged 4 weeks to <2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 4 weeks to <2 years of age. Cohort 1 (6 months - <2 years): Subjects must be <2 years of age at the Week 2 visit therefore the maximum age at screening is 22 months.

Cohort 2 (4 weeks - <6 months): Subjects must be <6 months of age at the Week 2 visit, therefore the maximum age at screening is 4 months for entry into this cohort.

* Parent or legal guardian is willing and able to provide written informed consent for the subject to participate in the trial.
* Screening plasma HIV-1 RNA level >=400copies/mL.
* Subjects who, in the investigator's opinion, and following viral resistance testing if conducted, are able to construct an active Nucleoside Reverse Transcriptase Inhibitor (NRTI) backbone regimen consisting of 2 NRTIs.
* Subjects must meet one of the following criteria:

Therapy-naïve or PI-naïve subjects (defined as having received less than one week of any PI).

PI-experienced subjects defined as having prior experience with no more than three PIs. Prior RTV-boosted PI therapy will be considered as only one PI as long as the RTV dose was lower than that recommended for use of RTV as an antiretroviral agent.

Exclusion Criteria:

* Prior history of having received APV.
* Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) therapy within 14 days prior to study drug administration (single or multiple dose) or anticipated need for concurrent NNRTI therapy during the study period.
* PI therapy within 5 days prior to study drug administration (applicable only for subjects undergoing single dose visits)
* Subjects and/or parents/legal guardians who, in the investigator's opinion, are not able to comply with the requirements of the study.
* Subject is in the initial acute phase of a Centers for Disease Control and Prevention (CDC) Clinical Category C event or infection (per 1994 classification) at Baseline. Subject may be enrolled provided they are receiving treatment for the infections, such treatment not being contraindicated with FPV, and subjects are clinically improving at the Baseline visit.
* Presence of a malabsorption syndrome or other gastrointestinal dysfunction which might interfere with drug absorption or render the subject unable to take oral medication.
* Presence of any serious medical condition (e.g., hemoglobinopathy, chronic anemia, diabetes, cardiac dysfunction, hepatitis, or clinically relevant pancreatitis) which, in the opinion of the investigator, might compromise the safety of the subject.
* Any acute laboratory abnormality at screen which, in the opinion of the investigator, should preclude the subject's participation in the study of an investigational compound. If subjects are found to have an acute Grade 4 laboratory abnormality at screening, this test may be repeated once within the screening window. Any verified Grade 4 laboratory abnormality would exclude a subject from study participation.
* Grade 3 or higher (>10x ULN) serum aminotransferase levels (alanine aminotransferase, ALT and/or aspartate aminotransferase, AST) within 28 days prior to study drug administration and / or clinically relevant hepatitis within the previous 6 months.
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days of study drug administration or an anticipated need for such treatment within the study period.
* Treatment with immunomodulating agents (e.g., systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (e.g., hydroxyurea or foscarnet) within 28 days of study drug administration.
* Treatment with any of the following medications within 28 days prior to receiving study medication or the anticipated need during the study:

Amiodarone, astemizole, bepridil, bupropion, cisapride, clorazepate, clozapine, diazepam, dihydroergotamine, encainide, ergonovine, ergotamine, estazolam, flecainide, flurazepam, lovastatin, meperidine, methylergonovine, midazolam, pimozide, piroxicam, propafenone, propoxyphene, quinidine, simvastatin, terfenadine, and triazolam (these drugs have been excluded for safety reasons).

Carbamazepine, dexamethasone, phenobarbital, primidone, rifampin, St Johns Wort, (these drugs have been excluded because they have the potential to decrease plasma protease inhibitor concentrations).

* Treatment with other investigational drugs/therapies within 28 days prior to receiving study medication (note: treatments available through a Treatment IND or other expanded-access mechanism will be evaluated on a case-by-case basis in consultation with the sponsor).
* History of drug or other allergy which, in the opinion of the investigator, contraindicates participation in the trial or known hypersensitivity to any study medications (e.g. documented hypersensitivity to a nucleoside analogue).

Ages: 4 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2003-10-23 (Actual); Primary Completion 2011-07-05 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (14):
- United States (2):
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Durham, North Carolina
- GSK Investigational Site, Buenos Aires, Argentina
- Mexico (2):
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- Portugal (3):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Lisbon
- GSK Investigational Site, San Juan, Puerto Rico
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Africa (3):
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Parow Valley, Western Province
  - GSK Investigational Site, Soweto

REFERENCES:
- [Background] Cotton M, Cassim H, Pavia-Ruz N, Garges HP, Perger T, Ford SL, Wire MB, Givens N, Ross LL, Lou Y, Sievers J, Cheng K. Pharmacokinetics, safety and antiviral activity of fosamprenavir/ritonavir-containing regimens in HIV-infected children aged 4 weeks to 2 years-48-week study data. Pediatr Infect Dis J. 2014 Jan;33(1):57-62. doi: 10.1097/INF.0b013e3182a1123a. PMID 23811743

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 23-Oct-2003 to 29-March-2022 in Argentina, Mexico, Portugal and South Africa. The cut off date for 48 week primary endpoint was July 5th 2011.
Pre-assignment Details: 59 participants were enrolled in the study and received at least one dose of Fosamprenavir (FPV)/Ritonavir (RTV) (Safety Population). Five participants out of 59 only received single dose before discontinuing the study. 54 participants who received both single and multiple doses of FPV/RTV were included in Intent to Treat-Exposed (ITT-E) population.
Groups:
- Cohort 1, Arm A - 6 Months to <2 Years: Participants with Human immunodeficiency virus (HIV-1) in Cohort 1 were initially administered single dose of fosamprenavir (FPV) 30 milligrams per kilogram (mg/kg) at single dose visit 1 (SDV1) or single dose of FPV/RTV 30/6 mg/kg (SDV2). Participants who underwent SDV2 administration began individualized regimens ranging from FPV 30 to 45/RTV 6 to 7 mg/kg twice a day (BID). Subsequently enrolled participants were administered with FPV/RTV 45/7 mg/kg BID.
- Cohort 2, Arm A - 4 Weeks to <6 Months: Participants with HIV-1 in Cohort 2 were initially administered with single dose administration of FPV/RTV 45/7 mg/kg (SDV1). The FPV/RTV dosage regimen selected for chronic dosing ranged from 30/7 mg/kg BID to 60/10 mg/kg BID. Subsequently enrolled participants were administered with FPV/RTV 45/10 mg/kg BID.
Period: Overall Study
Arm/Group | Cohort 1, Arm A - 6 Months to <2 Years | Cohort 2, Arm A - 4 Weeks to <6 Months
Started | 28 | 26
Completed | 21 | 18
Not Completed | 7 | 8
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 0 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Insufficient Viral Load Response | 1 | 1
Not completed — Lack of availability of RTV | 1 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Relocation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received both single and multiple doses of FPV/RTV were included in Intent to Treat-Exposed (ITT-E) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Arm A - 6 Months to <2 Years | Cohort 2, Arm A - 4 Weeks to <6 Months | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.3 (5.6) | 3.4 (0.95) | 8.6 (6.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 0 | 9
  Not Hispanic or Latino | 19 | 26 | 45
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Plasma Amprenavir (APV) AUC (0-tau[τ])
Description: Plasma samples were assayed for APV concentrations using a validated assay. The GlaxoSmithKline (GSK) Department of Clinical Pharmacology Modeling and Simulation conducted pharmacokinetic (PK) analysis of the plasma APV concentration-time data using a model-independent approach. As a measure of total drug exposure, the area under the plasma-concentration-versus-time curve over the dosing interval at steady-state (AUC[0-τ]), where "τ" is the length of the dosing interval, was calculated by the linear up/log down trapezoidal method. hours, hr.
Time Frame: Week 48
Population: Pharmacokinetic (PK) Population: all participants for whom serial plasma PK samples were analyzed. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hr per microgram/milliliter (hr*µg/mL)
Groups:
- FPV/RTV BID: 4 Weeks to <6 Months: Participants initially underwent two single dose visits (SDV): 30 milligrams per kilogram (mg/kg) fosamprenavir (FPV) oral suspension, 30/6 mg/kg FPV/ritonavir (RTV) oral solution, followed by individualized dosing (30/7 mg/kg BID to 60/10 mg/kg FPV/RTV twice a day [BID]). Per data for Cohort 1, participants in Cohort 2 underwent one SDV (45/7 mg/kg FPV/RTV), followed by individualized dosing (30/7 mg/kg to 60/10 mg/kg FPV/RTV BID). Additional enrolled participants in Cohort 2 later received 45/10 mg/kg FPV/RTV BID.
- FPV/RTV BID: 6 Months to <2 Years: Participants initially underwent two single dose visits (SDV): 30 milligrams per kilogram (mg/kg) fosamprenavir (FPV) oral suspension, 30/6 mg/kg FPV/ritonavir (RTV) oral solution, followed by individualized dosing (30/7 mg/kg BID to 60/10 mg/kg FPV/RTV twice a day [BID]). Per preliminary data at Week 2, the chronic dosing regimen for Cohort 1 was 45/7 mg/kg FPV/RTV BID, then changed to 45/7 mg/kg FPV/RTV BID with an increase to 60/7 mg/kg FPV/RTV BID at Week 2; later, per another analysis, all additional participants enrolled remained on 45/7 mg/kg FPV/RTV BID throughout.
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 9 | 10
Hr per microgram/milliliter (hr*µg/mL)
  45/10 mg/kg BID; n=9, 1: number analyzed (Participants) | 9 | 1
  45/10 mg/kg BID; n=9, 1 | 26.6 [15.2 to 46.8] | 64.51 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 1.
  60/10 mg/kg BID; n=2, 2: number analyzed (Participants) | 2 | 2
  60/10 mg/kg BID; n=2, 2 | 54.2 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 26.22 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2.
  45/7 mg/kg BID; n=2, 10: number analyzed (Participants) | 2 | 10
  45/7 mg/kg BID; n=2, 10 | 35.08 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 27.5 [14.5 to 52.1]
  60/7 mg/kg BID; n=0, 8: number analyzed (Participants) | 0 | 8
  60/7 mg/kg BID; n=0, 8 |  | 48.4 [12.9 to 181.5]

2. Primary Outcome: Plasma APV Cmax
Description: The maximum concentration at steady state (Cmax) was measured.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Micrograms per milliliter (µg/mL)
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 9 | 10
Micrograms per milliliter (µg/mL)
  45/10 mg/kg BID; n=9, 1: number analyzed (Participants) | 9 | 1
  45/10 mg/kg BID; n=9, 1 | 6.25 [3.82 to 10.2] | 21.82 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 1.
  60/10 mg/kg BID; n=2, 2: number analyzed (Participants) | 2 | 2
  60/10 mg/kg BID; n=2, 2 | 10.44 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 7.47 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2.
  45/7 mg/kg BID; n=2, 10: number analyzed (Participants) | 2 | 10
  45/7 mg/kg BID; n=2, 10 | 8.20 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 5.84 [3.35 to 10.2]
  60/7 mg/kg BID; n=0, 9: number analyzed (Participants) | 0 | 9
  60/7 mg/kg BID; n=0, 9 |  | 10.4 [3.64 to 30.0]

3. Primary Outcome: Plasma APV Cτ
Description: The plasma concentration at the end of the dosing interval at steady state (Cτ) was measured.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter (µg/mL)
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 11 | 29
Micrograms per milliliter (µg/mL)
  45/10 mg/kg BID; n=11, 15: number analyzed (Participants) | 11 | 15
  45/10 mg/kg BID; n=11, 15 | 0.86 [0.50 to 1.48] | 1.92 [1.42 to 2.58]
  60/10 mg/kg BID; n=3, 5: number analyzed (Participants) | 3 | 5
  60/10 mg/kg BID; n=3, 5 | 0.60 [NA to 127.50] — Because of the small sample size, the lower limit of the confidence interval cannot be reliably calculated. | 2.58 [1.29 to 5.17]
  45/7 mg/kg BID; n=3, 29: number analyzed (Participants) | 3 | 29
  45/7 mg/kg BID; n=3, 29 | 0.44 [0.18 to 1.07] | 2.17 [1.69 to 2.80]
  60/7 mg/kg BID; n=0, 12: number analyzed (Participants) | 0 | 12
  60/7 mg/kg BID; n=0, 12 |  | 2.81 [1.69 to 4.67]

4. Primary Outcome: Plasma APV CL/F Following Dosing Expressed in mL/Min/kg
Description: Apparent clearance of drug from plasma following extravascular administration (CL/F) was calculated using the formulation: APV Dose in mg/kg units divided by AUC(0-τ). For FPV, doses were expressed in APV molar equivalents (50 mg of FPV = 43.2 mg of APV). Normalizing CL/F for bodyweight allows for comparison of CL/F across populations.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters/minute/kilogram (mL/min/kg)
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 9 | 10
Milliliters/minute/kilogram (mL/min/kg)
  45/10 mg/kg BID; n=9, 1: number analyzed (Participants) | 9 | 1
  45/10 mg/kg BID; n=9, 1 | 22.9 [12.9 to 40.6] | 10.42 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 1.
  60/10 mg/kg BID; n=2, 2: number analyzed (Participants) | 2 | 2
  60/10 mg/kg BID; n=2, 2 | 15.3 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 31.92 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2.
  45/7 mg/kg BID; n=2, 10: number analyzed (Participants) | 2 | 10
  45/7 mg/kg BID; n=2, 10 | 17.50 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 22.8 [12.0 to 43.1]
  60/7 mg/kg BID; n=0, 8: number analyzed (Participants) | 0 | 8
  60/7 mg/kg BID; n=0, 8 |  | 17.8 [4.75 to 66.7]

5. Primary Outcome: Plasma APV CL/F Following Dosing Expressed in mL/Min
Description: Apparent clearance of drug from plasma following extravascular administration (CL/F) was calculated as dose/AUC(0-τ). For FPV, doses were expressed in APV molar equivalents (50 mg of FPV = 43.2 mg of APV).
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 9 | 10
mL/min
  45/10 mg/kg BID; n=9, 1: number analyzed (Participants) | 9 | 1
  45/10 mg/kg BID; n=9, 1 | 135 [69.1 to 262] | 62.5 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 1.
  60/10 mg/kg BID; n=2, 2: number analyzed (Participants) | 2 | 2
  60/10 mg/kg BID; n=2, 2 | 86.4 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 234.3 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2.
  45/7 mg/kg BID; n=2, 10: number analyzed (Participants) | 2 | 10
  45/7 mg/kg BID; n=2, 10 | 106.7 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 190 [93.2 to 386.2]
  60/7 mg/kg BID; n=0, 8: number analyzed (Participants) | 0 | 8
  60/7 mg/kg BID; n=0, 8 |  | 172 [46.3 to 638]

6. Primary Outcome: Plasma Unbound APV Cτ
Description: Participants who are <2 years old may have reduced protein binding; therefore, plasma unbound APV concentrations were measured to determine dosing recommendations at acceptable dosing volumes. Unbound or "free" APV is the fraction of drug that is not bound to protein. Cτ is the plasma concentration at the end of the dosing interval at steady state.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 7 | 16
µg/mL
  45/10 mg/kg BID; n=7, 16 | 0.091 (0.083) | 0.087 (0.076)
  60/10 mg/kg BID; n=1, 7: number analyzed (Participants) | 1 | 7
  60/10 mg/kg BID; n=1, 7 | 0.003 (NA) — The standard deviation is not available because the number of participants analyzed is 1. | 0.069 (0.052)
  45/7 mg/kg BID; n=1, 16: number analyzed (Participants) | 1 | 16
  45/7 mg/kg BID; n=1, 16 | 0.027 (NA) — The standard deviation is not available because the number of participants analyzed is 1. | 0.150 (0.086)
  60/7 mg/kg BID; n=0, 12: number analyzed (Participants) | 0 | 12
  60/7 mg/kg BID; n=0, 12 |  | 0.290 (0.310)

7. Primary Outcome: Plasma Unbound APV Percent Protein Binding (%Cτ)
Description: Participants who are <2 years old may have reduced protein binding; therefore, plasma unbound APV concentrations were measured to determine dosing recommendations at acceptable dosing volumes. APV %Cτ unbound is the percentage of the total APV Cτ that is unbound.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of total APV Cτ unbound
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 7 | 16
Percentage of total APV Cτ unbound
  45/10 mg/kg BID; n=7, 15: number analyzed (Participants) | 7 | 15
  45/10 mg/kg BID; n=7, 15 | 5.79 (2.05) | 6.56 (2.27)
  60/10 mg/kg BID; n=1, 7: number analyzed (Participants) | 1 | 7
  60/10 mg/kg BID; n=1, 7 | 5.32 (NA) — The standard deviation is not available because the number of participants analyzed is 1. | 5.81 (1.68)
  45/7 mg/kg BID; n=1, 16: number analyzed (Participants) | 1 | 16
  45/7 mg/kg BID; n=1, 16 | 7.55 (NA) — The standard deviation is not available because the number of participants analyzed is 1. | 8.23 (8.67)
  60/7 mg/kg BID; n=0, 9: number analyzed (Participants) | 0 | 9
  60/7 mg/kg BID; n=0, 9 |  | 9.20 (5.39)

8. Primary Outcome: Absolute Values of Alanine Amino Transferase (ALT) and Aspartate Amino Transferase (AST) at Baseline (Day 1), Weeks 4, 12, 24, 36, and 48
Description: Blood samples of the participants were collected for the evaluation of ALT and AST. Clinical chemistry analyses were carried out using the observed analysis strategy.
Time Frame: Baseline (Day 1) and Weeks 4, 12, 24, 36, and 48
Population: Safety Population: all participants with documented evidence of having received at least one dose of investigational treatment. Only those participants contributing data were analyzed.
Measure: Median (Inter-Quartile Range); unit: International units per liter (IU/L)
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 26 | 30
International units per liter (IU/L)
  ALT, Day 1; n=26;30 | 22.0 [6 to 94] | 20.0 [9 to 884]
  ALT, Week 4; n=23;28: number analyzed (Participants) | 23 | 28
  ALT, Week 4; n=23;28 | 14.0 [6 to 25] | 15.5 [8 to 164]
  ALT, Week 12; n=22;27: number analyzed (Participants) | 22 | 27
  ALT, Week 12; n=22;27 | 15.0 [8 to 35] | 15.0 [8 to 39]
  ALT, Week 24; n=22;26: number analyzed (Participants) | 22 | 26
  ALT, Week 24; n=22;26 | 16.0 [7 to 37] | 15.5 [4 to 111]
  ALT, Week 36; n=20;25: number analyzed (Participants) | 20 | 25
  ALT, Week 36; n=20;25 | 15.5 [10 to 51] | 16.0 [8 to 134]
  ALT, Week 48; n=18;24: number analyzed (Participants) | 18 | 24
  ALT, Week 48; n=18;24 | 15.0 [7 to 42] | 16.0 [9 to 36]
  AST, Day 1; n=26;30 | 43.5 [24 to 165] | 44.0 [29 to 852]
  AST, Week 4; n=23;28: number analyzed (Participants) | 23 | 28
  AST, Week 4; n=23;28 | 32.0 [21 to 49] | 35.0 [23 to 150]
  AST, Week 12; n=22;27: number analyzed (Participants) | 22 | 27
  AST, Week 12; n=22;27 | 35.0 [21 to 63] | 40.0 [23 to 67]
  AST, Week 24; n=22;26: number analyzed (Participants) | 22 | 26
  AST, Week 24; n=22;26 | 34.0 [25 to 43] | 36.5 [17 to 109]
  AST, Week 36; n=20;24: number analyzed (Participants) | 20 | 24
  AST, Week 36; n=20;24 | 35.0 [21 to 58] | 34.0 [22 to 105]
  AST, Week 48; n=18;23: number analyzed (Participants) | 18 | 23
  AST, Week 48; n=18;23 | 34.5 [17 to 58] | 34.0 [22 to 57]

9. Primary Outcome: Absolute Values of Cholesterol, Glucose, High Density Lipoprotein (HDL) Cholesterol, Low Density Lipoprotein (LDL) and Triglyceride (TG) at Baseline (Day 1), Weeks 4, 12, 24, 36, and 48
Description: Blood samples of all participants were generally collected under non-fasting conditions (given the age of participants) for the evaluation of cholesterol, serum glucose, HDL cholesterol, LDL cholesterol and triglyceride (TG). Clinical chemistry analyses were carried out using the observed analysis strategy.
Time Frame: Baseline (Day 1) and Weeks 4, 12, 24, 36, and 48
Population: Safety Population. Only those participants contributing data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Millimoles per liter (mmol/L)
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 26 | 30
Millimoles per liter (mmol/L)
  Cholesterol, Day 1; n=22;29: number analyzed (Participants) | 22 | 29
  Cholesterol, Day 1; n=22;29 | 2.235 [1.900 to 2.780] | 2.910 [2.640 to 3.530]
  Cholesterol, Week 4; n=4;2: number analyzed (Participants) | 4 | 2
  Cholesterol, Week 4; n=4;2 | 3.085 [2.430 to 3.180] | 3.885 [3.220 to 4.550]
  Cholesterol, Week 12; n=0;2: number analyzed (Participants) | 0 | 2
  Cholesterol, Week 12; n=0;2 |  | 3.950 [3.300 to 4.550]
  Cholesterol, Week 24; n=22;26: number analyzed (Participants) | 22 | 26
  Cholesterol, Week 24; n=22;26 | 4.175 [3.300 to 5.210] | 4.000 [3.490 to 5.050]
  Cholesterol, Week 36; n=3;2: number analyzed (Participants) | 3 | 2
  Cholesterol, Week 36; n=3;2 | 3.030 [1.600 to 3.390] | 3.150 [2.900 to 3.400]
  Cholesterol, Week 48; n=18;24: number analyzed (Participants) | 18 | 24
  Cholesterol, Week 48; n=18;24 | 3.890 [3.270 to 4.700] | 4.750 [3.850 to 5.285]
  Glucose, Day 1; n=26;30 | 4.80 [4.50 to 5.20] | 4.70 [4.40 to 5.20]
  Glucose, Week 4; n=23;28: number analyzed (Participants) | 23 | 28
  Glucose, Week 4; n=23;28 | 4.60 [4.30 to 5.30] | 4.80 [4.20 to 5.20]
  Glucose, Week 12; n=22;27: number analyzed (Participants) | 22 | 27
  Glucose, Week 12; n=22;27 | 4.70 [4.10 to 5.50] | 4.70 [4.30 to 5.30]
  Glucose, Week 24; n=22;26: number analyzed (Participants) | 22 | 26
  Glucose, Week 24; n=22;26 | 4.55 [4.00 to 4.90] | 4.30 [4.00 to 5.00]
  Glucose, Week 36; n=20;25: number analyzed (Participants) | 20 | 25
  Glucose, Week 36; n=20;25 | 4.50 [4.35 to 5.10] | 4.60 [4.30 to 4.80]
  Glucose, Week 48; n=18;24: number analyzed (Participants) | 18 | 24
  Glucose, Week 48; n=18;24 | 4.45 [4.20 to 4.90] | 4.70 [4.35 to 5.15]
  HDL, Day 1; n=22;29: number analyzed (Participants) | 22 | 29
  HDL, Day 1; n=22;29 | 0.655 [0.410 to 0.810] | 0.680 [0.500 to 0.850]
  HDL, Week 4; n=4;2: number analyzed (Participants) | 4 | 2
  HDL, Week 4; n=4;2 | 0.825 [0.585 to 0.970] | 0.690 [0.650 to 0.730]
  HDL, Week 12; n=0;2: number analyzed (Participants) | 0 | 2
  HDL, Week 12; n=0;2 |  | 0.775 [0.650 to 0.900]
  HDL, Week 24; n=22;26: number analyzed (Participants) | 22 | 26
  HDL, Week 24; n=22;26 | 0.900 [0.720 to 1.000] | 0.960 [0.800 to 1.100]
  HDL, Week 36; n=3;2: number analyzed (Participants) | 3 | 2
  HDL, Week 36; n=3;2 | 0.640 [0.400 to 0.700] | 0.805 [0.610 to 1.000]
  HDL, Week 48; n=18;24: number analyzed (Participants) | 18 | 24
  HDL, Week 48; n=18;24 | 0.825 [0.730 to 1.000] | 1.050 [0.805 to 1.200]
  LDL, Day 1; n=22;28: number analyzed (Participants) | 22 | 28
  LDL, Day 1; n=22;28 | 0.90 [0.65 to 1.15] | 1.50 [1.11 to 1.94]
  LDL, Week 4; n=4;2: number analyzed (Participants) | 4 | 2
  LDL, Week 4; n=4;2 | 1.25 [0.85 to 1.48] | 2.45 [1.90 to 3.00]
  LDL, Week 12; n=0;2: number analyzed (Participants) | 0 | 2
  LDL, Week 12; n=0;2 |  | 2.33 [2.00 to 2.66]
  LDL, Week 24; n=22;26: number analyzed (Participants) | 22 | 26
  LDL, Week 24; n=22;26 | 2.08 [1.10 to 3.10] | 2.32 [2.00 to 3.10]
  LDL, Week 36; n=3;2: number analyzed (Participants) | 3 | 2
  LDL, Week 36; n=3;2 | 1.90 [0.30 to 2.10] | 2.08 [1.75 to 2.40]
  LDL, Week 48; n=18;24: number analyzed (Participants) | 18 | 24
  LDL, Week 48; n=18;24 | 2.33 [1.70 to 2.85] | 2.80 [2.50 to 3.37]
  TG, Day 1; n=22;29: number analyzed (Participants) | 22 | 29
  TG, Day 1; n=22;29 | 1.695 [1.220 to 2.280] | 1.650 [1.300 to 2.100]
  TG, Week 4; n=4;2: number analyzed (Participants) | 4 | 2
  TG, Week 4; n=4;2 | 2.015 [1.505 to 2.280] | 1.645 [1.310 to 1.980]
  TG, Week 12; n=0;2: number analyzed (Participants) | 0 | 2
  TG, Week 12; n=0;2 |  | 1.810 [0.800 to 2.820]
  TG, Week 24; n=22;26: number analyzed (Participants) | 22 | 26
  TG, Week 24; n=22;26 | 2.155 [1.580 to 2.710] | 1.550 [1.100 to 2.120]
  TG, Week 36; n=3;2: number analyzed (Participants) | 3 | 2
  TG, Week 36; n=3;2 | 1.310 [1.100 to 2.000] | 1.700 [1.100 to 2.300]
  TG, Week 48; n=18;24: number analyzed (Participants) | 18 | 24
  TG, Week 48; n=18;24 | 1.590 [1.270 to 2.010] | 1.390 [0.920 to 1.950]

10. Primary Outcome: Absolute Values of Serum Lipase at Baseline (Day 1), Weeks 4, 12, 24, and 48
Description: Blood samples of all participants were collected for the evaluation of serum lipase. Clinical chemistry analyses were carried out using the observed analysis strategy. Change from Baseline in serum lipase was calculated as the value at the indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1) and Weeks 4, 12, 24, and 48
Population: Safety Population. Only those participants contributing data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Units per liter (U/L)
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 2 | 11
Units per liter (U/L)
  Day 1; n=2;11 | 20.5 [20.0 to 21.0] | 22.0 [17.0 to 38.0]
  Week 4; n=0;1: number analyzed (Participants) | 0 | 1
  Week 4; n=0;1 |  | 16.0 [16.0 to 16.0]
  Week 12; n=0;1: number analyzed (Participants) | 0 | 1
  Week 12; n=0;1 |  | 68.0 [68.0 to 68.0]
  Week 24; n=0;8: number analyzed (Participants) | 0 | 8
  Week 24; n=0;8 |  | 19.5 [14.5 to 28.0]
  Week 48; n=1;8: number analyzed (Participants) | 1 | 8
  Week 48; n=1;8 | 16.0 [16.0 to 16.0] | 16.0 [14.5 to 24.0]

11. Primary Outcome: Number of Participants With the Indicated Treatment-emergent (TE) Grade 3/4 Laboratory Abnormalities
Description: TE toxicities were presented for each laboratory parameter. A toxicity was considered TE if it was greater than the Baseline grade, and if it was observed on/after the date of the first dose of study drug (SD), and on/before the date of the last dose of SD. Per the Division of AIDS Table for Grading the Severity of Adult and Pediatric AEs, Grade 3=severe; Grade 4=potentially life-threatening.
Time Frame: Baseline (Day 1) until Week 48
Population: Safety Population. Only those participants contributing data were analyzed.
Measure: Number; unit: participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 29 | 30
participants
  Clinical Chemistry Toxicities - Grade 3 | 2 | 4
  Clinical Chemistry Toxicities - Grade 4 | 0 | 1
  Hematology Toxicities - Grade 3 | 2 | 2
  Hematology Toxicities - Grade 4 | 0 | 1

12. Primary Outcome: Number of Participants With the Indicated Treatment-emergent (TE) Grade 3/4 Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE is considered TE if it has an onset date on or after the date of the first dose of study drug, and on or before the date of the final dose of study drug. As per the Division of AIDS Table for Grading the Severity of Adult and Pediatric AEs, Grade 3=severe; Grade 4=potentially life-threatening.
Time Frame: Baseline (Day 1) until Week 48
Population: Safety Population. In addition to the 54 participants starting FPV/RTV BID treatment, the FPV/RTV BID treatment group includes 5 participants who only received investigational product at the single dose visits in APV20002.
Measure: Number; unit: participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 29 | 30
participants | 11 | 10

13. Primary Outcome: Number of Participants Who Permanently Discontinued the Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline (Day 1) until Week 48
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 29 | 30
participants | 1 | 2

14. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (that could include a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Day 1 and up to week 684
Population: Safety population included participants receiving FPV or FPV/RTV at any dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 29 | 30
Participants | 25 | 29

15. Other Pre Specified Outcome: Number of Participants With Clinical Chemistry Toxicities
Description: Blood samples were collected for the analysis of all clinical chemistry parameters. Laboratory toxicities were graded using the Division of AIDS (DAIDS) table for grading the severity of adult and pediatric adverse events, where grade 1=mild, grade 2=moderate, grade 3=severe and grade 4=potentially life-threatening. Results for participants with Grade 1 to 4 clinical chemistry toxicities is presented.
Time Frame: Day 1 and up to Week 684
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 29 | 30
Participants
  Grade 1 | 5 | 5
  Grade 2 | 9 | 14
  Grade 3 | 3 | 7
  Grade 4 | 1 | 1

16. Other Pre Specified Outcome: Number of Participants With Hematology Toxicities
Description: Blood samples were collected for the analysis of all hematology parameters. Laboratory toxicities were graded using the DAIDS Table for grading the severity of adult and pediatric adverse events, where grade 1=mild, grade 2=moderate, grade 3=severe and grade 4=potentially life-threatening. Results for participants with Grade 1 to 4 hematology toxicities is presented.
Time Frame: Day 1 and up to Week 684
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 29 | 30
Participants
  Grade 1 | 6 | 6
  Grade 2 | 5 | 6
  Grade 3 | 3 | 2
  Grade 4 | 0 | 2

17. Other Pre Specified Outcome: Number of Participants With Treatment Limiting Toxicities
Description: Treatment limiting toxicities are defined as those that are related to investigational medicinal products and deemed to be unacceptable, leading to restriction of further dose escalation.
Time Frame: Day 1 and up to Week 684
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 29 | 30
Participants | 0 | 0

18. Other Pre Specified Outcome: Number of Participants Who Permanently Discontinued the Treatment Due to Adverse Event
Description: as for outcome 14
Time Frame: Day 1 and up to Week 684
Population: Intent-to-Treat exposed
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 29 | 30
Participants | 1 | 1

19. Secondary Outcome: Number of Participants With Plasma Human Immuno Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Levels < 400 Copies/Milliliter at Each Study Visit
Description: Blood samples of participants were collected to measure plasma HIV-1 RNA concentrations.
Time Frame: Baseline (Day 1) and up to Week 684
Population: Intent to treat- exposed (ITT-E) Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 26 | 28
Participants
  Baseline (Day 1) | 1 | 0
  Week 4: number analyzed (Participants) | 21 | 28
  Week 4 | 5 | 6
  Week 12: number analyzed (Participants) | 22 | 27
  Week 12 | 13 | 18
  Week 24: number analyzed (Participants) | 22 | 25
  Week 24 | 18 | 20
  Week 36: number analyzed (Participants) | 21 | 25
  Week 36 | 19 | 20
  Week 48: number analyzed (Participants) | 18 | 24
  Week 48 | 15 | 22
  Week 60: number analyzed (Participants) | 16 | 16
  Week 60 | 15 | 12
  Week 72: number analyzed (Participants) | 16 | 15
  Week 72 | 14 | 14
  Week 84: number analyzed (Participants) | 16 | 16
  Week 84 | 14 | 15
  Week 96: number analyzed (Participants) | 15 | 14
  Week 96 | 15 | 14
  Week 108: number analyzed (Participants) | 15 | 14
  Week 108 | 15 | 14
  Week 120: number analyzed (Participants) | 14 | 12
  Week 120 | 14 | 11
  Week 132: number analyzed (Participants) | 14 | 11
  Week 132 | 14 | 11
  Week 144: number analyzed (Participants) | 14 | 9
  Week 144 | 14 | 8
  Week 156: number analyzed (Participants) | 14 | 10
  Week 156 | 14 | 10
  Week 168: number analyzed (Participants) | 12 | 9
  Week 168 | 12 | 9
  Week 180: number analyzed (Participants) | 10 | 9
  Week 180 | 10 | 9
  Week 192: number analyzed (Participants) | 10 | 8
  Week 192 | 10 | 8
  Week 204: number analyzed (Participants) | 10 | 9
  Week 204 | 10 | 9
  Week 216: number analyzed (Participants) | 11 | 9
  Week 216 | 10 | 9
  Week 228: number analyzed (Participants) | 12 | 8
  Week 228 | 12 | 8
  Week 240: number analyzed (Participants) | 12 | 8
  Week 240 | 12 | 8
  Week 252: number analyzed (Participants) | 12 | 8
  Week 252 | 12 | 8
  Week 264: number analyzed (Participants) | 12 | 8
  Week 264 | 12 | 8
  Week 276: number analyzed (Participants) | 12 | 8
  Week 276 | 12 | 8
  Week 288: number analyzed (Participants) | 12 | 8
  Week 288 | 12 | 8
  Week 300: number analyzed (Participants) | 12 | 8
  Week 300 | 12 | 8
  Week 312: number analyzed (Participants) | 12 | 8
  Week 312 | 10 | 8
  Week 324: number analyzed (Participants) | 11 | 8
  Week 324 | 11 | 8
  Week 336: number analyzed (Participants) | 11 | 7
  Week 336 | 11 | 7
  Week 348: number analyzed (Participants) | 10 | 6
  Week 348 | 10 | 6
  Week 360: number analyzed (Participants) | 11 | 7
  Week 360 | 10 | 7
  Week 372: number analyzed (Participants) | 11 | 7
  Week 372 | 11 | 7
  Week 384: number analyzed (Participants) | 11 | 7
  Week 384 | 10 | 7
  Week 396: number analyzed (Participants) | 11 | 7
  Week 396 | 11 | 7
  Week 408: number analyzed (Participants) | 11 | 7
  Week 408 | 11 | 7
  Week 420: number analyzed (Participants) | 9 | 7
  Week 420 | 8 | 7
  Week 432: number analyzed (Participants) | 10 | 7
  Week 432 | 10 | 7
  Week 444: number analyzed (Participants) | 10 | 7
  Week 444 | 9 | 7
  Week 456: number analyzed (Participants) | 9 | 7
  Week 456 | 9 | 7
  Week 468: number analyzed (Participants) | 9 | 7
  Week 468 | 9 | 7
  Week 480: number analyzed (Participants) | 9 | 7
  Week 480 | 9 | 7
  Week 492: number analyzed (Participants) | 8 | 7
  Week 492 | 7 | 7
  Week 504: number analyzed (Participants) | 9 | 7
  Week 504 | 9 | 7
  Week 516: number analyzed (Participants) | 9 | 7
  Week 516 | 9 | 7
  Week 528: number analyzed (Participants) | 9 | 6
  Week 528 | 9 | 6
  Week 540: number analyzed (Participants) | 9 | 5
  Week 540 | 9 | 5
  Week 552: number analyzed (Participants) | 9 | 5
  Week 552 | 9 | 5
  Week 564: number analyzed (Participants) | 6 | 5
  Week 564 | 6 | 5
  Week 576: number analyzed (Participants) | 6 | 5
  Week 576 | 6 | 5
  Week 588: number analyzed (Participants) | 6 | 5
  Week 588 | 6 | 5
  Week 600: number analyzed (Participants) | 6 | 3
  Week 600 | 5 | 3
  Week 612: number analyzed (Participants) | 5 | 3
  Week 612 | 5 | 3
  Week 624: number analyzed (Participants) | 5 | 3
  Week 624 | 5 | 3
  Week 636: number analyzed (Participants) | 1 | 2
  Week 636 | 1 | 2
  Week 648: number analyzed (Participants) | 1 | 2
  Week 648 | 1 | 2
  Week 660: number analyzed (Participants) | 1 | 2
  Week 660 | 1 | 2
  Week 672: number analyzed (Participants) | 0 | 2
  Week 672 | 0 | 2
  Week 684: number analyzed (Participants) | 0 | 1
  Week 684 | 0 | 1

20. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA Levels at Each Study Visit
Description: Blood samples of participants were collected to measure plasma HIV-1 RNA copies. Baseline value was defined as the value observed at the day 1 visit or if this value is missing the last value observed before the start of investigational product. Change from baseline value was defined as post-dose value minus baseline value.
Time Frame: Baseline (Day 1) and up to Week 684
Population: Intent to treat-exposed (ITT-E) Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Log10 copies/milliliter
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 22 | 28
Log10 copies/milliliter
  Week 4: number analyzed (Participants) | 21 | 28
  Week 4 | -2.38 [-2.89 to -1.64] | -2.33 [-2.87 to -1.95]
  Week 12: number analyzed (Participants) | 22 | 27
  Week 12 | -3.11 [-3.94 to -1.91] | -3.14 [-3.58 to -2.12]
  Week 24: number analyzed (Participants) | 22 | 25
  Week 24 | -3.77 [-4.21 to -1.91] | -3.38 [-3.88 to -2.39]
  Week 36: number analyzed (Participants) | 21 | 25
  Week 36 | -3.72 [-4.26 to -3.00] | -3.52 [-3.90 to -2.69]
  Week 48: number analyzed (Participants) | 18 | 24
  Week 48 | -3.90 [-4.48 to -2.28] | -3.56 [-3.92 to -3.12]
  Week 60: number analyzed (Participants) | 16 | 16
  Week 60 | -3.89 [-4.63 to -2.45] | -3.12 [-3.92 to -2.04]
  Week 72: number analyzed (Participants) | 16 | 15
  Week 72 | -3.95 [-4.63 to -2.45] | -3.60 [-3.93 to -2.69]
  Week 84: number analyzed (Participants) | 16 | 16
  Week 84 | -3.95 [-4.63 to -3.11] | -3.62 [-3.98 to -2.97]
  Week 96: number analyzed (Participants) | 15 | 14
  Week 96 | -4.26 [-4.71 to -3.31] | -3.70 [-3.93 to -3.00]
  Week 108: number analyzed (Participants) | 15 | 14
  Week 108 | -4.26 [-4.71 to -3.31] | -3.80 [-3.93 to -3.00]
  Week 120: number analyzed (Participants) | 14 | 12
  Week 120 | -4.12 [-4.71 to -3.31] | -3.58 [-3.90 to -2.82]
  Week 132: number analyzed (Participants) | 14 | 11
  Week 132 | -4.09 [-4.71 to -3.31] | -3.52 [-3.90 to -2.80]
  Week 144: number analyzed (Participants) | 14 | 9
  Week 144 | -4.12 [-4.71 to -3.31] | -3.52 [-3.90 to -2.95]
  Week 156: number analyzed (Participants) | 14 | 10
  Week 156 | -4.12 [-4.71 to -3.31] | -3.34 [-3.90 to -2.95]
  Week 168: number analyzed (Participants) | 12 | 9
  Week 168 | -3.95 [-4.63 to -3.15] | -3.52 [-3.90 to -2.95]
  Week 180: number analyzed (Participants) | 10 | 9
  Week 180 | -4.36 [-4.71 to -3.90] | -3.52 [-3.90 to -2.95]
  Week 192: number analyzed (Participants) | 10 | 8
  Week 192 | -4.28 [-4.71 to -3.90] | -3.31 [-3.90 to -2.87]
  Week 204: number analyzed (Participants) | 10 | 9
  Week 204 | -4.22 [-4.71 to -3.00] | -3.52 [-3.99 to -2.95]
  Week 216: number analyzed (Participants) | 11 | 9
  Week 216 | -4.36 [-4.71 to -3.00] | -3.52 [-3.99 to -2.95]
  Week 228: number analyzed (Participants) | 12 | 8
  Week 228 | -4.45 [-4.85 to -3.46] | -3.71 [-4.06 to -3.07]
  Week 240: number analyzed (Participants) | 12 | 8
  Week 240 | -4.22 [-4.64 to -3.46] | -3.71 [-4.06 to -3.07]
  Week 252: number analyzed (Participants) | 12 | 8
  Week 252 | -4.22 [-4.64 to -3.46] | -3.71 [-4.06 to -3.07]
  Week 264: number analyzed (Participants) | 12 | 8
  Week 264 | -4.22 [-4.64 to -3.46] | -3.71 [-4.06 to -3.07]
  Week 276: number analyzed (Participants) | 12 | 8
  Week 276 | -4.22 [-4.64 to -3.46] | -3.71 [-4.06 to -3.07]
  Week 288: number analyzed (Participants) | 12 | 8
  Week 288 | -4.22 [-4.64 to -3.56] | -3.71 [-4.06 to -2.94]
  Week 300: number analyzed (Participants) | 12 | 8
  Week 300 | -4.22 [-4.64 to -3.56] | -3.80 [-4.07 to -3.29]
  Week 312: number analyzed (Participants) | 12 | 8
  Week 312 | -4.05 [-4.61 to -2.25] | -3.98 [-4.07 to -3.36]
  Week 324: number analyzed (Participants) | 11 | 8
  Week 324 | -4.01 [-4.65 to -3.10] | -3.87 [-4.07 to -3.36]
  Week 336: number analyzed (Participants) | 11 | 7
  Week 336 | -4.09 [-4.81 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 348: number analyzed (Participants) | 10 | 6
  Week 348 | -4.33 [-4.81 to -3.10] | -3.36 [-3.99 to -3.05]
  Week 360: number analyzed (Participants) | 11 | 7
  Week 360 | -4.09 [-4.81 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 372: number analyzed (Participants) | 11 | 7
  Week 372 | -4.09 [-4.81 to -3.10] | -3.36 [-4.13 to -2.79]
  Week 384: number analyzed (Participants) | 11 | 7
  Week 384 | -4.01 [-4.65 to -3.10] | -3.15 [-4.13 to -3.05]
  Week 396: number analyzed (Participants) | 11 | 7
  Week 396 | -4.09 [-4.81 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 408: number analyzed (Participants) | 11 | 7
  Week 408 | -4.09 [-4.81 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 420: number analyzed (Participants) | 9 | 7
  Week 420 | -4.09 [-4.65 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 432: number analyzed (Participants) | 10 | 7
  Week 432 | -4.33 [-4.81 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 444: number analyzed (Participants) | 10 | 7
  Week 444 | -4.04 [-4.65 to -2.64] | -3.62 [-4.13 to -3.05]
  Week 456: number analyzed (Participants) | 9 | 7
  Week 456 | -4.09 [-4.65 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 468: number analyzed (Participants) | 9 | 7
  Week 468 | -4.09 [-4.65 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 480: number analyzed (Participants) | 9 | 7
  Week 480 | -4.09 [-4.65 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 492: number analyzed (Participants) | 8 | 7
  Week 492 | -3.55 [-4.61 to -2.50] | -3.62 [-4.13 to -3.05]
  Week 504: number analyzed (Participants) | 9 | 7
  Week 504 | -4.09 [-4.65 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 516: number analyzed (Participants) | 9 | 7
  Week 516 | -4.09 [-4.65 to -3.10] | -3.62 [-4.13 to -3.05]
  Week 528: number analyzed (Participants) | 9 | 6
  Week 528 | -4.09 [-4.65 to -3.10] | -3.80 [-4.13 to -3.05]
  Week 540: number analyzed (Participants) | 9 | 5
  Week 540 | -4.09 [-4.65 to -3.10] | -3.99 [-4.13 to -3.62]
  Week 552: number analyzed (Participants) | 9 | 5
  Week 552 | -4.09 [-4.65 to -3.10] | -3.99 [-4.13 to -3.62]
  Week 564: number analyzed (Participants) | 6 | 5
  Week 564 | -4.28 [-4.65 to -3.10] | -3.99 [-4.13 to -3.62]
  Week 576: number analyzed (Participants) | 6 | 5
  Week 576 | -4.04 [-4.65 to -3.10] | -3.99 [-4.13 to -3.62]
  Week 588: number analyzed (Participants) | 6 | 5
  Week 588 | -4.04 [-4.65 to -3.10] | -3.99 [-4.13 to -3.62]
  Week 600: number analyzed (Participants) | 6 | 3
  Week 600 | -3.55 [-4.09 to -1.53] | -3.99 [-4.56 to -3.62]
  Week 612: number analyzed (Participants) | 5 | 3
  Week 612 | -4.09 [-4.65 to -4.00] | -3.99 [-4.56 to -3.62]
  Week 624: number analyzed (Participants) | 5 | 3
  Week 624 | -4.09 [-4.65 to -4.00] | -3.99 [-4.56 to -3.62]
  Week 636: number analyzed (Participants) | 1 | 2
  Week 636 | -4.00 [-4.99 to -4.00] | -4.27 [-4.56 to -3.99]
  Week 648: number analyzed (Participants) | 1 | 2
  Week 648 | -4.00 [-4.00 to -4.00] | -4.27 [-4.56 to -3.99]
  Week 660: number analyzed (Participants) | 1 | 2
  Week 660 | -4.09 [-4.09 to -4.09] | -4.27 [-4.56 to -3.99]
  Week 672: number analyzed (Participants) | 0 | 2
  Week 672 |  | -4.27 [-4.56 to -3.99]
  Week 684: number analyzed (Participants) | 0 | 1
  Week 684 |  | -3.99 [-3.99 to -3.99]

21. Secondary Outcome: Absolute Values of Cluster of Differentiation 4 (CD4+) Cell Counts by Study Visit
Description: Blood samples of participants were collected for the measurement of the CD4+ cells.
Time Frame: Baseline (Day 1) and up to week 684
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: Cells/cubic millimeter
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 23 | 28
Cells/cubic millimeter
  Baseline (Day 1) | 1378 [950 to 1690] | 1120 [873.5 to 1827.5]
  Week 4 | 1610 [1170 to 2520] | 1734.5 [1290 to 2287]
  Week 12: number analyzed (Participants) | 22 | 27
  Week 12 | 1405 [1107 to 1757] | 1822 [1120 to 2392]
  Week 24: number analyzed (Participants) | 22 | 26
  Week 24 | 1595 [1320 to 1910] | 1475.5 [1223 to 2178]
  Week 36: number analyzed (Participants) | 21 | 25
  Week 36 | 1780 [1620 to 2410] | 1523 [1200 to 2069]
  Week 48: number analyzed (Participants) | 17 | 24
  Week 48 | 1690 [1150 to 2080] | 1602 [1035 to 2345.5]
  Week 60: number analyzed (Participants) | 15 | 16
  Week 60 | 1890 [1544 to 1980] | 1311 [944 to 1962]
  Week 72: number analyzed (Participants) | 15 | 15
  Week 72 | 1407 [1172 to 1890] | 1667 [930 to 1883]
  Week 84: number analyzed (Participants) | 15 | 16
  Week 84 | 1560 [1280 to 2044] | 1490.5 [1307.5 to 2516.5]
  Week 96: number analyzed (Participants) | 15 | 13
  Week 96 | 1530 [1055 to 1990] | 1460 [1260 to 1730]
  Week 108: number analyzed (Participants) | 15 | 14
  Week 108 | 1440 [1220 to 1820] | 1343.5 [1149 to 1610]
  Week 120: number analyzed (Participants) | 14 | 12
  Week 120 | 1480 [1160 to 1940] | 1148.5 [905.5 to 1735]
  Week 132: number analyzed (Participants) | 14 | 10
  Week 132 | 1285 [1130 to 1430] | 1440 [1033 to 1810]
  Week 144: number analyzed (Participants) | 14 | 10
  Week 144 | 1250 [935 to 1480] | 1562 [1141 to 1730]
  Week 156: number analyzed (Participants) | 14 | 10
  Week 156 | 1422 [990 to 1600] | 1307 [1147 to 1719]
  Week 168: number analyzed (Participants) | 13 | 9
  Week 168 | 1550 [1150 to 1700] | 1236 [883 to 1358]
  Week 180: number analyzed (Participants) | 12 | 9
  Week 180 | 1331.5 [983 to 1700] | 978 [939 to 1640]
  Week 192: number analyzed (Participants) | 12 | 9
  Week 192 | 1339 [944.5 to 1644] | 1327 [877 to 1559]
  Week 204: number analyzed (Participants) | 12 | 9
  Week 204 | 1160 [776.5 to 1690] | 1082 [960 to 1650]
  Week 216: number analyzed (Participants) | 12 | 9
  Week 216 | 1336 [979.5 to 1451.5] | 909 [809 to 1497]
  Week 228: number analyzed (Participants) | 12 | 8
  Week 228 | 1136 [910.5 to 1345] | 1106 [842 to 1425]
  Week 240: number analyzed (Participants) | 12 | 8
  Week 240 | 1132.5 [736.5 to 1464] | 1067 [743.5 to 1232.5]
  Week 252: number analyzed (Participants) | 12 | 8
  Week 252 | 1379 [927 to 1592] | 1098.5 [796 to 1454]
  Week 264: number analyzed (Participants) | 11 | 8
  Week 264 | 1109 [990 to 1326] | 853 [777 to 1421.5]
  Week 276: number analyzed (Participants) | 12 | 8
  Week 276 | 1180.5 [889.5 to 1336] | 970 [803.5 to 1238]
  Week 288: number analyzed (Participants) | 12 | 8
  Week 288 | 1063 [737.5 to 1330] | 911.5 [832 to 1140.5]
  Week 300: number analyzed (Participants) | 12 | 8
  Week 300 | 1062 [659 to 1249] | 990 [571.5 to 1188.5]
  Week 312: number analyzed (Participants) | 12 | 8
  Week 312 | 924 [775 to 1199.5] | 928.5 [858 to 1220]
  Week 324: number analyzed (Participants) | 11 | 8
  Week 324 | 980 [770 to 1310] | 1242 [840.4 to 1420]
  Week 336: number analyzed (Participants) | 11 | 7
  Week 336 | 856 [670 to 1160] | 1160 [711 to 1276]
  Week 348: number analyzed (Participants) | 11 | 7
  Week 348 | 1030 [840 to 1365] | 976 [887 to 1264]
  Week 360: number analyzed (Participants) | 10 | 7
  Week 360 | 1151 [839 to 1240] | 962 [759 to 1310]
  Week 372: number analyzed (Participants) | 11 | 7
  Week 372 | 1051 [700 to 1070] | 926 [637 to 1545]
  Week 384: number analyzed (Participants) | 10 | 7
  Week 384 | 950 [800 to 1158] | 884 [731 to 1281]
  Week 396: number analyzed (Participants) | 10 | 7
  Week 396 | 971 [805 to 1110] | 900 [630 to 1148]
  Week 408: number analyzed (Participants) | 10 | 6
  Week 408 | 1005 [770 to 1107] | 938.5 [578 to 1106]
  Week 420: number analyzed (Participants) | 9 | 7
  Week 420 | 840 [768 to 1130] | 850 [705 to 1007]
  Week 432: number analyzed (Participants) | 8 | 7
  Week 432 | 940.5 [705 to 1138] | 918 [754 to 1121]
  Week 444: number analyzed (Participants) | 8 | 7
  Week 444 | 811 [745.5 to 990] | 860 [816 to 1139]
  Week 456: number analyzed (Participants) | 9 | 7
  Week 456 | 1003 [712 to 1143] | 832 [701 to 1080]
  Week 468: number analyzed (Participants) | 8 | 6
  Week 468 | 910 [665 to 1211] | 863 [715 to 1024]
  Week 480: number analyzed (Participants) | 6 | 6
  Week 480 | 1063.5 [838 to 1270] | 1010 [760 to 1226]
  Week 492: number analyzed (Participants) | 9 | 7
  Week 492 | 839 [780 to 970] | 930 [823 to 1139]
  Week 504: number analyzed (Participants) | 9 | 7
  Week 504 | 887 [805 to 1013] | 910 [777 to 1265]
  Week 516: number analyzed (Participants) | 8 | 7
  Week 516 | 776 [699.5 to 952] | 994 [793 to 1121]
  Week 528: number analyzed (Participants) | 9 | 7
  Week 528 | 860 [690 to 1070] | 892 [732 to 1136]
  Week 540: number analyzed (Participants) | 9 | 5
  Week 540 | 851 [720 to 976] | 877 [798 to 1040]
  Week 552: number analyzed (Participants) | 9 | 5
  Week 552 | 756 [730 to 940] | 1000 [941 to 1080]
  Week 564: number analyzed (Participants) | 7 | 5
  Week 564 | 908 [809 to 1110] | 804 [790 to 890]
  Week 576: number analyzed (Participants) | 6 | 5
  Week 576 | 792 [768 to 1013] | 990 [910 to 1047]
  Week 588: number analyzed (Participants) | 6 | 5
  Week 588 | 873 [750 to 1018] | 1100 [870 to 1110]
  Week 600: number analyzed (Participants) | 6 | 2
  Week 600 | 865.5 [813 to 936] | 717 [506 to 928]
  Week 612: number analyzed (Participants) | 5 | 3
  Week 612 | 720 [714 to 800] | 949 [655 to 1000]
  Week 624: number analyzed (Participants) | 4 | 3
  Week 624 | 753 [678.5 to 884.5] | 720 [500 to 1020]
  Week 636: number analyzed (Participants) | 2 | 2
  Week 636 | 770 [610 to 930] | 535 [290 to 580]
  Week 648: number analyzed (Participants) | 2 | 2
  Week 648 | 720 [660 to 780] | 455 [450 to 460]
  Week 660: number analyzed (Participants) | 1 | 2
  Week 660 | 750 [750 to 750] | 610 [320 to 900]
  Week 672: number analyzed (Participants) | 0 | 2
  Week 672 |  | 710 [490 to 930]
  Week 684: number analyzed (Participants) | 0 | 1
  Week 684 |  | 580 [580 to 580]

22. Secondary Outcome: Plasma FPV Concentrations
Time Frame: Post -Week 48 through Week 684
Population: All PK data collected through 5 July 2011 were included in the 48-week analysis results, no data was subsequently collected.
Groups:
- FPV/RTV BID: Participants with Human immunodeficiency virus (HIV-1) of age group-6 months to <2 years were administered with fosamprenavir (FPV)/ritonavir (RTV) 45/7 milligrams per kilogram (mg/kg) twice a day (BID) and participants with HIV-1 of age group - 4 weeks to <6 months were administered with FPV/RTV 45/10 mg/kg BID. FPV/RTV BID arm also include participants who only received treatment at single dose visits (SDV).
Arm/Group | FPV/RTV BID
Number analyzed (Participants) | 0

23. Secondary Outcome: Number of Participants With Treatment-Emergent Mutations at Virologic Failure Timepoint
Description: A blood sample was drawn from participants failing to respond to therapy, and genotyping was performed to identify the mutations present in the baseline (pre-therapy) and the sample obtained at virologic failure (VF). For each participant, the HIV-1 mutations found at the time of failure were compared with any HIV-1 mutations detected in the blood sample at baseline. New International AIDS Society-USA defined resistance mutations that developed at the time of failure were tabulated by drug class- NRTI, nucleoside reverse transcriptase inhibitor; NNRTI, non-nucleoside reverse transcriptase inhibitor; PI, protease inhibitor. Participants are grouped by study arm (prior therapy experience), results displayed in this table are from participants who met virologic failure criteria from Week 48 through Week 684.
Time Frame: Week 48 to Week 684
Population: VF population included participants who failed to achieve plasma HIV-RNA<400 copies/mL by Week 24; or confirmed HIV-RNA rebound to >=400 copies/mL any time after achieving plasma HIV-RNA<400 copies/mL and had evaluable viral isolate genotypic data. Only participants with an HIV-1 genotype which obtained for both the baseline and the indicated time of VF points were evaluable. No participants in this time frame were PI-experienced, therefore data was not collected for the PI-Experienced Group.
Measure: Count of Participants; unit: Participants
Groups:
- ART-Naive: Antiretroviral therapy (ART) Naive participants with HIV-1 of age group-6 months to <2 years were administered with FPV/RTV 45/7 mg/kg BID and participants with HIV-1 of age group - 4 weeks to <6 months were administered with FPV/RTV 45/10 mg/kg BID.
- PI-Naive: PI-Naive participants with HIV-1 of age group-6 months to <2 years were administered with FPV/RTV 45/7 mg/kg BID and participants with HIV-1 of age group - 4 weeks to <6 months were administered with FPV/RTV 45/10 mg/kg BID.
- PI-Experienced: PI-Experienced participants with HIV-1 of age group-6 months to <2 years were administered with FPV/RTV 45/7 mg/kg BID and participants with HIV-1 of age group - 4 weeks to <6 months were administered with FPV/RTV 45/10 mg/kg BID.
Arm/Group | ART-Naive | PI-Naive | PI-Experienced
Number analyzed (Participants) | 1 | 2 | 0
Participants
  PRO, L10L/R | 1 | 0 |
  PRO, I62I/V | 1 | 0 |

24. Secondary Outcome: Number of Participants With Treatment-Emergent Changes in HIV-1 Phenotypic Drug Susceptibility
Description: A blood sample was drawn from participant failing to respond to therapy, and the mutations present in the virus were identified. Phenotypic resistance was assessed for virologic failure population and evaluated for Protease Inhibitors (PIs), Nucleotide reverse transcriptase inhibitors (NRTIs), and non-NRTIs (NNTRIs) using Monogram PhenoSense Assay. Virologic failure was defined as having failed to achieve a plasma HIV-RNA of <400 copies/mL by Week 24 or having had a confirmed HIV-RNA rebound to ≥400 c/mL at any time after achieving a plasma HIV-RNA of <400 c/mL.
Time Frame: Post-Week 48 to Week 684
Population: Virological failure population includes participants who met the protocol definition of definition of virologic failure and for whom an HIV-1 phenotype was obtained at both the baseline (pre-therapy) and at the virologic failure timepoints. No participants in this time frame were PI-experienced, therefore data was not collected for the PI-Experienced Arm/Group.
Measure: Count of Participants; unit: Participants
Arm/Group | ART-Naive | PI-Naive | PI-Experienced
Number analyzed (Participants) | 1 | 2 | 0
Participants
  Treatment emergent reduced NRTI drug susceptibility | 0 | 0 |
  Treatment emergent reduced NNRTI drug susceptibility | 0 | 0 |
  Treatment emergent reduced PI drug susceptibility | 0 | 0 |

25. Secondary Outcome: Number of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) <400 Copies Per Milliliter at Baseline and Weeks 4, 12, 24, 36, and 48 (MSD=F)
Description: Blood samples of participants were collected to measure plasma HIV-1 RNA concentrations. Viral load, measured in RNA copies per milliliter of plasma, is an efficacy measure for antiretroviral drugs. In the Missing, Switch, or Discontinuation=Failure (MSD=F) analysis, participants who had missing data at or had discontinued the study prior to a certain time point or had changed their background antiretroviral regimen are classified as non-responders.
Time Frame: Baseline and Weeks 4, 12, 24, 36, and 48
Population: Intent-to-Treat Exposed (ITT-E) Population: participants who received chronic therapy with FPV or FPV/RTV at any dose. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 26 | 28
participants
  Baseline | 1 | 0
  Week 4: number analyzed (Participants) | 21 | 28
  Week 4 | 5 | 6
  Week 12: number analyzed (Participants) | 22 | 27
  Week 12 | 13 | 18
  Week 24: number analyzed (Participants) | 22 | 25
  Week 24 | 18 | 20
  Week 36: number analyzed (Participants) | 21 | 25
  Week 36 | 19 | 20
  Week 48: number analyzed (Participants) | 18 | 24
  Week 48 | 15 | 22

26. Secondary Outcome: Median Plasma HIV-1 RNA (log10 Copies/mL) at Baseline and Weeks 4, 12, 24, 36, and 48 (Observed Analysis)
Description: Blood samples of participants were collected to assess the decrease in the number of HIV-1 RNA copies.
Time Frame: Baseline and Weeks 4, 12, 24, 36, and 48
Population: ITT-E Population. In the observed analysis, data are presented for the number of participants still enrolled in the study at a certain time point.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 26 | 28
log10 copies/mL
  Baseline, n=26;28 | 5.80 [5.17 to 6.30] | 5.51 [4.81 to 5.76]
  Week 4, n=21;28: number analyzed (Participants) | 21 | 28
  Week 4, n=21;28 | 3.29 [2.88 to 4.05] | 2.88 [2.65 to 3.19]
  Week 12, n=22;27: number analyzed (Participants) | 22 | 27
  Week 12, n=22;27 | 2.28 [1.69 to 3.11] | 2.07 [1.69 to 2.72]
  Week 24, n=22;25: number analyzed (Participants) | 22 | 25
  Week 24, n=22;25 | 1.69 [1.69 to 2.27] | 1.74 [1.69 to 2.34]
  Week 36, n=21;25: number analyzed (Participants) | 21 | 25
  Week 36, n=21;25 | 1.69 [1.69 to 2.33] | 1.69 [1.69 to 1.80]
  Week 48, n=18;24: number analyzed (Participants) | 18 | 24
  Week 48, n=18;24 | 1.69 [1.69 to 1.69] | 1.69 [1.69 to 1.72]

27. Secondary Outcome: Median Change From Baseline in Plasma HIV-1 RNA (log10 Copies/mL) at Weeks 4, 12, 24, 36, and 48 (Observed Analysis)
Description: Blood samples of participants were collected to assess the decrease in the number of HIV-1 RNA copies. Change from Baseline in plasma HIV-1 RNA was calculated as the value at the indicated time point minus the value at Baseline.
Time Frame: Baseline and Weeks 4, 12, 24, 36, and 48
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 26 | 28
log10 copies/mL
  Week 4, n=21;28: number analyzed (Participants) | 21 | 28
  Week 4, n=21;28 | -2.38 [-2.89 to -1.64] | -2.33 [-2.87 to -1.95]
  Week 12, n=22;27: number analyzed (Participants) | 22 | 27
  Week 12, n=22;27 | -3.11 [-3.94 to -1.94] | -3.14 [-3.58 to -2.12]
  Week 24, n=22;25: number analyzed (Participants) | 22 | 25
  Week 24, n=22;25 | -3.77 [-4.21 to -1.91] | -3.38 [-3.88 to -2.39]
  Week 36, n=21;25: number analyzed (Participants) | 21 | 25
  Week 36, n=21;25 | -3.72 [-4.26 to -3.00] | -3.52 [-3.90 to -2.69]
  Week 48, n=18;24: number analyzed (Participants) | 18 | 24
  Week 48, n=18;24 | -3.90 [-4.48 to -2.28] | -3.56 [-3.92 to -3.12]

28. Secondary Outcome: Number of Participants With at Least a 1.0 log10 HIV-1 RNA Decrease From Baseline at Weeks 4, 12, 24, 36, and 48 (MSD=F Analysis)
Description: Blood samples of participants were collected to assess the decrease in the number of HIV-1 RNA copies. In the MSD=F analysis, participants who had missing data at or had discontinued the study prior to a certain time point or had changed their background antiretroviral regimen are classified as non-responders.
Time Frame: Baseline and Weeks 4, 12, 24, 36, and 48
Population: ITT-E Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 26 | 28
participants
  Week 4 | 16 | 25
  Week 12 | 21 | 25
  Week 24 | 21 | 23
  Week 36 | 19 | 22
  Week 48 | 16 | 21

29. Secondary Outcome: Median Percent Cluster of Differentiation Antigen 4 (CD4+) Cell Count at Baseline and at Weeks 4, 12, 24, 36, and 48
Description: Blood samples of participants were collected for the measurement of the percentage of total lymphocytes that are CD4+ cells. Observed analysis was used for the summary of proportion endpoints using viral load data. CD4+ cells are white blood cells that are important in fighting infection. HIV infects CD4+ cells, replicates in them, and destroys them. A CD4+ cell count provides a measure of the status of the immune system and to what extent it is affected by HIV.
Time Frame: Baseline and Weeks 4, 12, 24, 36, and 48
Population: ITT-E Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percentage of cells
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 23 | 28
Percentage of cells
  Baseline, n=23;28 | 27 [20 to 36] | 25 [18 to 31]
  Week 4, n=23;28 | 29 [23 to 37] | 27.5 [20.5 to 35]
  Week 12, n=22;27: number analyzed (Participants) | 22 | 27
  Week 12, n=22;27 | 27.5 [23.6 to 35] | 32 [23 to 39.4]
  Week 24, n=22;26: number analyzed (Participants) | 22 | 26
  Week 24, n=22;26 | 31.5 [27.2 to 34] | 32.8 [26 to 37.7]
  Week 36, n=21;25: number analyzed (Participants) | 21 | 25
  Week 36, n=21;25 | 32 [26 to 38.8] | 29.5 [28 to 36.5]
  Week 48, n=18;24: number analyzed (Participants) | 18 | 24
  Week 48, n=18;24 | 28 [25 to 32] | 31.6 [23 to 38]

30. Secondary Outcome: Median Percent Change From Baseline in CD4+ Cell Count at Weeks 4, 12, 24, 36, and 48
Description: Blood samples of participants were collected for the measurement of the percentage of total lymphocytes that are CD4+ cells. Observed analysis was used for the summary of proportion endpoints using viral load data. Change from Baseline in percentage was calculated as the value at indicated time points minus the value at Baseline.
Time Frame: Baseline and Weeks 4, 12, 24, 36, and 48
Population: ITT-E Population. Only those participants contributing data at the indicated time points were analyzed. Not all participants had values at both baseline and the indicated time points; thus, change from baseline could not be calculated for all participants.
Measure: Median (Inter-Quartile Range); unit: Percentage of cells
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 20 | 28
Percentage of cells
  Week 4, n=20;28 | 3 [-1 to 7.5] | 3.4 [0 to 6.3]
  Week 12, n=19;27: number analyzed (Participants) | 19 | 27
  Week 12, n=19;27 | 2 [0 to 8] | 6 [2 to 8]
  Week 24, n=19;26: number analyzed (Participants) | 19 | 26
  Week 24, n=19;26 | 7 [-1 to 12] | 6 [2.6 to 11]
  Week 36, n=18;25: number analyzed (Participants) | 18 | 25
  Week 36, n=18;25 | 8 [3 to 12] | 5 [3 to 8]
  Week 48, n=15;24: number analyzed (Participants) | 15 | 24
  Week 48, n=15;24 | 5 [-7 to 9] | 4.7 [2.2 to 8.7]

31. Secondary Outcome: Number of Participants With the Indicated Virological Outcome at Week 48
Description: Blood samples of participants were collected to measure plasma HIV-1 RNA concentrations. PI-exp = PI-experienced. Virologic success was defined as plasma HIV-1 RNA <400 copies/mL. Virologic failure: (1) HIV-1 RNA >=400 copies/mL, (2) change of background antiretroviral treatment (ART), (3) discontinued study due to lack of efficacy, (4) discontinued study with last HIV-1 >=400 copies/mL. No virologic data at Week 48 window: (a) discontinued study due to an adverse event or death, (b) discontinued study due to other reasons (withdrew consent, loss to follow-up, moved, etc.).
Time Frame: Week 48
Population: ITT-E Population. Only those participants contributing data were analyzed.
Measure: Number; unit: participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 26 | 28
participants
  Virological (V) success | 15 | 20
  V failure (1) | 3 | 2
  V failure (2) | 0 | 2
  V failure (3) | 1 | 1
  V failure (4) | 2 | 1
  No V data at Week 48 (a) | 1 | 1
  No V data at Week 48 (b) | 4 | 1

32. Secondary Outcome: Plasma Ritonavir (RTV) AUC (0-τ)
Description: Plasma samples were assayed for RTV concentrations using a validated assay. The GSK Department of Clinical Pharmacology Modeling and Simulation conducted PK analysis of the plasma RTV concentration-time data using a model-independent approach. As a measure of total drug exposure, the area under the plasma-concentration-versus-time curve over the dosing interval at steady-state (AUC[0-τ]), where τ is the length of the dosing interval, was calculated by the linear up/log down trapezoidal method.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*µg/mL
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 11 | 22
hr*µg/mL
  7 mg/kg BID; n=2, 22: number analyzed (Participants) | 2 | 22
  7 mg/kg BID; n=2, 22 | 1.921 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 7.363 [4.769 to 11.369]
  10 mg/kg BID; n=11, 2: number analyzed (Participants) | 11 | 2
  10 mg/kg BID; n=11, 2 | 12.952 [6.932 to 24.200] | 18.750 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2.

33. Secondary Outcome: Plasma RTV Cmax
Description: The maximum concentration at steady state (Cmax) was measured.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 12 | 23
µg/mL
  7 mg/kg BID, n=2, 23: number analyzed (Participants) | 2 | 23
  7 mg/kg BID, n=2, 23 | 0.404 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 1.576 [0.991 to 2.506]
  10 mg/kg BID, n=12, 2: number analyzed (Participants) | 12 | 2
  10 mg/kg BID, n=12, 2 | 2.388 [1.364 to 4.180] | 3.823 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2.

34. Secondary Outcome: Plasma RTV Cτ
Description: The plasma concentration at the end of the dosing interval at steady state (Cτ) was measured.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 15 | 33
µg/mL
  7 mg/kg BID, n=4, 33: number analyzed (Participants) | 4 | 33
  7 mg/kg BID, n=4, 33 | 0.0795 [0.0316 to 0.1996] | 0.2468 [0.1875 to 0.3249]
  10 mg/kg BID, n=15, 19: number analyzed (Participants) | 15 | 19
  10 mg/kg BID, n=15, 19 | 0.1855 [0.1146 to 0.3003] | 0.4200 [0.2958 to 0.5962]

35. Secondary Outcome: Plasma RTV CL/F Expressed in mL/Min/kg
Description: Apparent clearance of drug from plasma following extravascular administration (CL/F) was calculated as dose in mg/kg units divided by AUC(0-τ). Normalizing CL/F for bodyweight allows for comparison of CL/F across populations.
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min/kg
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 11 | 22
mL/min/kg
  7 mg/kg BID, n=2, 22: number analyzed (Participants) | 2 | 22
  7 mg/kg BID, n=2, 22 | 58.668 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 14.960 [9.762 to 22.927]
  10 mg/kg BID, n=11, 2: number analyzed (Participants) | 11 | 2
  10 mg/kg BID, n=11, 2 | 12.118 [6.435 to 22.818] | 8.938 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2.

36. Secondary Outcome: Plasma RTV CL/F Expressed in mL/Min
Description: Apparent clearance of drug from plasma following extravascular administration (CL/F) was calculated as dose in mg/kg units divided by AUC(0-τ).
Time Frame: Week 48
Population: PK Population. Only those participants contributing data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 11 | 22
mL/min
  7 mg/kg BID, n=2, 22: number analyzed (Participants) | 2 | 22
  7 mg/kg BID, n=2, 22 | 335.2 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2. | 134.1 [87.3 to 205.8]
  10 mg/kg BID, n=11, 2: number analyzed (Participants) | 11 | 2
  10 mg/kg BID, n=11, 2 | 72.1 [38.7 to 134.3] | 57.9 [NA to NA] — The 95% CI is not available because the number of participants analyzed is 2.

37. Secondary Outcome: Number of Confirmed Virologic Failure Participants (Par.) With Treatment-emergent HIV Genotypic Resistance in Reverse Transcriptase and Protease
Description: A blood sample was drawn for par. failing to respond to therapy, and the mutations present in the virus were identified. For each par., the mutations found at the time of failure were compared with any mutations found in the blood sample at baseline. New International AIDS Society-USA defined resistance mutations that developed at the time of failure were tabulated by drug class. VF, virologic failure; NRTI, nucleoside reverse transcriptase inhibitor; NNRTI, non-nucleoside reverse transcriptase inhibitor; PI, protease inhibitor. Par. are grouped by study arm and prior therapy experience.
Time Frame: Baseline through Week 48
Population: VF: par. with failure to achieve plasma HIV-RNA <400 copies/mL by Week 24; or confirmed HIV-RNA rebound to >=400 copies/mL any time after achieving plasma HIV-RNA <400 copies/mL and had evaluable viral isolate genotypic and/or phenotypic data. Only par. contributing viral genotype at both baseline and the indicated time of VF points were evaluable.
Measure: Number; unit: participants
Groups:
- ART-naïve FPV/RTV Treatment Group: ART-naïve Human immunodeficiency virus (HIV)-1-infected pediatric participants (received no antiretroviral agents prior to study enrollment) were enrolled in one of two cohorts based on their age: 6 months to <2 years (Cohort 1); 4 weeks to <6 months (Cohort 2). Participants initially underwent single dose visits (SDV). Cohort 1: SDV 1: 30 milligrams per kilogram (mg/kg) fosamprenavir (FPV) oral suspension, followed by SDV 2: 30/6 mg/kg FPV/ritonavir (RTV) oral solution. Cohort 2: SDV 1: 45/7 mg/kg FPV/RTV. The chronic dosing regimen for Cohort 1 was 45/7 mg/kg twice a day (BID) FPV/RTV, and for Cohort 2 was 30/7 mg/kg BID to 60/10 mg/kg BID. Per the preliminary data at Week 2 in Cohort 1, additional enrolled participants received 60/7 mg/kg FPV/RTV BID; later, per another analysis, all additional participants enrolled remained on 45/7 mg/kg FPV/RTV BID with no dose increase at Week 2. In Cohort 2, additional enrolled participants received 45/10 mg/kg FPV/RTV BID.
- PI-naïve, ART-experienced FPV/RTV Treatment Group: PI-naïve, ART experienced, HIV-1-infected pediatric participants (received ART previously, but received <1 week's treatment with a PI) were enrolled in one of two cohorts based on their age: 6 months to <2 years (Cohort 1); 4 weeks to <6 months (Cohort 2). Participants initially underwent single dose visits (SDV). Cohort 1: SDV 1: 30 milligrams per kilogram (mg/kg) fosamprenavir (FPV) oral suspension, followed by SDV 2: 30/6 mg/kg FPV/ritonavir (RTV) oral solution. Cohort 2: SDV 1: 45/7 mg/kg FPV/RTV. The chronic dosing regimen for Cohort 1 was 45/7 mg/kg twice a day (BID) FPV/RTV, and for Cohort 2 was 30/7 mg/kg BID to 60/10 mg/kg BID. Per the preliminary data at Week 2 in Cohort 1, additional enrolled participants received 60/7 mg/kg FPV/RTV BID; later, per another analysis, all additional participants enrolled remained on 45/7 mg/kg FPV/RTV BID with no dose increase at Week 2. In Cohort 2, additional enrolled participants received 45/10 mg/kg FPV/RTV BID.
- PI-experienced, ART-experienced FPV/RTV Treatment Group: PI- experienced, ART-experienced, HIV-1-infected pediatric participants (received ART previously, and >1 week prior PI therapy [no more than 3 PIs before study enrollment]) were enrolled in one of two cohorts based on their age: 6 months to <2 years (Cohort 1); 4 weeks to <6 months (Cohort 2). Participants initially underwent SDVs. Cohort 1: SDV 1: 30 mg/kg fosamprenavir (FPV) oral suspension, followed by SDV 2: 30/6 mg/kg FPV/ritonavir (RTV) oral solution. Cohort 2: SDV 1: 45/7 mg/kg FPV/RTV. The chronic dosing regimen for Cohort 1 was 45/7 mg/kg twice a day (BID) FPV/RTV, and for Cohort 2 was 30/7 mg/kg BID to 60/10 mg/kg BID. Per the preliminary data at Week 2 in Cohort 1, additional enrolled participants received 60/7 mg/kg FPV/RTV BID; later, per another analysis, all additional participants enrolled remained on 45/7 mg/kg FPV/RTV BID with no dose increase at Week 2. In Cohort 2, additional enrolled participants received 45/10 mg/kg FPV/RTV BID.
Arm/Group | ART-naïve FPV/RTV Treatment Group | PI-naïve, ART-experienced FPV/RTV Treatment Group | PI-experienced, ART-experienced FPV/RTV Treatment Group
Number analyzed (Participants) | 2 | 3 | 2
participants
  Any HIV NRTI Mutation | 1 | 0 | 0
  HIV NRTI mutation M184V | 1 | 0 | 0
  Any HIV NNRTI Mutation | 0 | 0 | 1
  HIV NNRTI Mutation K101K/E | 0 | 0 | 1
  Any HIV Major PI Mutations | 0 | 0 | 0
  Any Minor HIV PI Mutations | 2 | 0 | 1
  Minor HIV PI Mutation L10F | 0 | 0 | 1
  Minor HIV PI Mutation L10I | 1 | 0 | 0
  Minor HIV PI Mutation L33L/F | 1 | 0 | 0
  Minor HIV PI Mutation L33F | 0 | 0 | 1

38. Secondary Outcome: Number of Confirmed Virologic Failure Participants (Par.) With Treatment-emergent Reductions in Drug Susceptibility (DS)
Description: A blood sample was drawn for par. failing to respond to therapy, and changes in DS for HIV isolated from the par. for each drug used in the study were assessed. The changes in DS detected by phenotypic assay in virus from the sample collected at the time of failure was compared with DS in the virus from the blood sample at baseline. Par. are grouped by study arm and prior therapy experience. DS is the state of HIV being susceptible to the antiretroviral agent (the virus can be inhibited by the drug). Reduced DS (i.e., HIV is resistant to the antiretroviral agent) can lead to treatment failure.
Time Frame: Baseline through Week 48
Population: VF: par. with failure to achieve plasma HIV-RNA <400 copies/mL by Week 24; or confirmed HIV-RNA rebound to >=400 copies/mL any time after achieving plasma HIV-RNA <400 copies/mL and had evaluable viral isolate genotypic and/or phenotypic data. Only par. contributing viral phenotype at both baseline and the indicated time of VF points were evaluable
Measure: Number; unit: participants
Groups:
- ART-experienced, PI-naïve FPV/RTV Treatment Group: PI-naïve, ART experienced, HIV-1-infected pediatric participants (received ART previously, but received <1 week's treatment with a PI) were enrolled in one of two cohorts based on their age: 6 months to <2 years (Cohort 1); 4 weeks to <6 months (Cohort 2). Participants initially underwent single dose visits (SDV). Cohort 1: SDV 1: 30 milligrams per kilogram (mg/kg) fosamprenavir (FPV) oral suspension, followed by SDV 2: 30/6 mg/kg FPV/ritonavir (RTV) oral solution. Cohort 2: SDV 1: 45/7 mg/kg FPV/RTV. The chronic dosing regimen for Cohort 1 was 45/7 mg/kg twice a day (BID) FPV/RTV, and for Cohort 2 was 30/7 mg/kg BID to 60/10 mg/kg BID. Per the preliminary data at Week 2 in Cohort 1, additional enrolled participants received 60/7 mg/kg FPV/RTV BID; later, per another analysis, all additional participants enrolled remained on 45/7 mg/kg FPV/RTV BID with no dose increase at Week 2. In Cohort 2, additional enrolled participants received 45/10 mg/kg FPV/RTV BID.
Arm/Group | ART-naïve FPV/RTV Treatment Group | ART-experienced, PI-naïve FPV/RTV Treatment Group | PI-experienced, ART-experienced FPV/RTV Treatment Group
Number analyzed (Participants) | 2 | 3 | 2
participants
  Any NRTI | 1 | 0 | 0
  Emtricitabine | 1 | 0 | 0
  Lamivudine | 1 | 0 | 0
  Any NNRTI | 0 | 0 | 0
  Any PI | 0 | 0 | 1
  Ritonavir-boosted Fosamprenavir | 0 | 0 | 1

39. Secondary Outcome: Number of Participants Reporting Perfect Adherence at Weeks 2, 12, 24, and 48 as Assessed by the Study Coordinator Using the Adherence Questionnaire
Description: A separate questionnaire was administered for FPV and RTV. Items 1-4 of the Adherence Questionnaire measured a participant's adherence with FPV or RTV during the last 3 days and the weekend prior to the indicated study visits. Perfect adherence was defined as not missing any doses of FPV or RTV since the last study visit.
Time Frame: Weeks 2, 12, 24, and 48
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 29 | 30
participants
  Week 2 | 18 | 24
  Week 12 | 17 | 24
  Week 24 | 19 | 21
  Week 48 | 13 | 17

40. Secondary Outcome: Number of Participants With the Indicated Response Scores for the Parent/Guardian (P/G) Perception of FPV Oral Suspension Questionnaire: Items 1 to 4
Description: P/G perceptions of FPV/RTV BID were assessed using a P/G Perception of Study Medication questionnaire administered during Weeks 2, 24, and 48/premature study discontinuation. Questions 1 to 4 ask directly about the P/G's assessment of 1=color, 2=texture/consistency, 3=odor, and 4=general satisfaction. Questions 5 to 10 ask about the P/G's perception of the child's assessment of the oral suspension. Data are reported as the number of participants with the indicated response by question, response category (1-3=dislike, 4=neutral, 5-7=like), and timing of visit.
Time Frame: Weeks 2, 24, and 48/premature study discontinuation
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 23 | 27
participants
  Week 2, color, dislike, n=23;27 | 3 | 5
  Week 2, color, neutral, n=23;27 | 7 | 13
  Week 2, color, like, n=23;27 | 13 | 9
  Week 24, color, dislike, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, color, dislike, n=20;24 | 4 | 4
  Week 24, color, neutral, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, color, neutral, n=20;24 | 2 | 10
  Week 24, color, like, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, color, like, n=20;24 | 14 | 10
  Week 48, color, dislike, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, color, dislike, n=15;22 | 6 | 7
  Week 48, color, neutral, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, color, neutral, n=15;22 | 1 | 7
  Week 48, color, like, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, color, like, n=15;22 | 8 | 8
  Week 2, texture, dislike, n=23;27 | 4 | 5
  Week 2, texture, neutral, n=23;27 | 7 | 10
  Week 2, texture, like, n=23;27 | 12 | 12
  Week 24, texture, dislike, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, texture, dislike, n=20;24 | 6 | 4
  Week 24, texture, neutral, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, texture, neutral, n=20;24 | 4 | 12
  Week 24, texture, like, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, texture, like, n=20;24 | 10 | 8
  Week 48, texture, dislike, n=15;21: number analyzed (Participants) | 15 | 21
  Week 48, texture, dislike, n=15;21 | 6 | 6
  Week 48, texture, neutral, n=15;21: number analyzed (Participants) | 15 | 21
  Week 48, texture, neutral, n=15;21 | 1 | 7
  Week 48, texture, like, n=15;21: number analyzed (Participants) | 15 | 21
  Week 48, texture, like, n=15;21 | 8 | 8
  Week 2, odor, dislike, n=23;27 | 1 | 7
  Week 2, odor, neutral, n=23;27 | 3 | 7
  Week 2, odor, like, n=23;27 | 19 | 13
  Week 24, odor, dislike, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, odor, dislike, n=20;24 | 4 | 7
  Week 24, odor, neutral, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, odor, neutral, n=20;24 | 2 | 8
  Week 24, odor, like, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, odor, like, n=20;24 | 14 | 9
  Week 48, odor, dislike, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, odor, dislike, n=15;22 | 4 | 7
  Week 48, odor, neutral, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, odor, neutral, n=15;22 | 1 | 5
  Week 48, odor, like, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, odor, like, n=15;22 | 10 | 10
  Week 2, general satisfaction, dislike, n=23;27 | 3 | 5
  Week 2, general satisfaction, neutral, n=23;27 | 4 | 7
  Week 2, general satisfaction, like, n=23;27 | 16 | 15
  Week 24, general satisfaction, dislike, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, general satisfaction, dislike, n=20;24 | 4 | 6
  Week 24, general satisfaction, neutral, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, general satisfaction, neutral, n=20;24 | 0 | 9
  Week 24, general satisfaction, like, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, general satisfaction, like, n=20;24 | 16 | 9
  Week 48, general satisfaction, dislike, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, general satisfaction, dislike, n=15;22 | 4 | 9
  Week 48, general satisfaction, neutral, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, general satisfaction, neutral, n=15;22 | 1 | 4
  Week 48, general satisfaction, like, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, general satisfaction, like, n=15;22 | 10 | 9

41. Secondary Outcome: Number of Participants With the Indicated Response Scores for the Parent/Guardian Perception of the Child's Assessment of FPV Oral Suspension Questionnaire: Items (I) 5 to 10
Description: Parent/guardian perceptions of FPV/RTV BID was assessed using a Parent/Guardian Perception of Study Medication questionnaire. Questions 1 to 4 ask directly about the parent/guardian's assessment of the color, texture/consistency, odor, and general satisfaction. Questions 5 to 10 ask about the parent/guardian's perception of the child's assessment of the oral suspension (Items: 5=reaction to new medicine [med.]; 6=taste; 7=acceptance; 8=swallowing; 9=willingness compared to other med.; 10=overall liking. Data for items 6/10 are reported in response categories: 1-3=dislike; 4=neutral; 5-7=like.
Time Frame: Weeks (W) 2, 24, and 48/premature study discontinuation
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
Number analyzed (Participants) | 23 | 27
participants
  W2, Item 5, takes all/most med. easily, n=23;27 | 10 | 11
  W2, Item 5, problem taking a few med., n=23;27 | 10 | 10
  W2, Item 5, problem taking most med., n=23;27 | 3 | 5
  W2, Item 5, impossible to take med., n=23;27 | 0 | 1
  W24, Item 5, takes all/most med. easily, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 5, takes all/most med. easily, n=20;23 | 12 | 10
  W24, Item 5, problem taking a few med., n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 5, problem taking a few med., n=20;23 | 8 | 7
  W24, Item 5, problem taking most med., n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 5, problem taking most med., n=20;23 | 0 | 5
  W24, Item 5, impossible to take med., n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 5, impossible to take med., n=20;23 | 0 | 1
  W48, Item 5, takes all/most med. easily, n=14;22: number analyzed (Participants) | 14 | 22
  W48, Item 5, takes all/most med. easily, n=14;22 | 10 | 17
  Week 48, Item 5, problem taking a few med., n=14;22: number analyzed (Participants) | 14 | 22
  Week 48, Item 5, problem taking a few med., n=14;22 | 4 | 5
  W48, Item 5, problem taking most med., n=14;22: number analyzed (Participants) | 14 | 22
  W48, Item 5, problem taking most med., n=14;22 | 0 | 0
  W48, Item 5, impossible to take med., n=14;22: number analyzed (Participants) | 14 | 22
  W48, Item 5, impossible to take med., n=14;22 | 0 | 0
  W2, Item 6, dislike, n=23;27 | 12 | 9
  W2, Item 6, neutral, n=23;27 | 4 | 10
  W2, Item 6, like, n=23;27 | 7 | 8
  W24, Item 6, dislike, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 6, dislike, n=20;23 | 11 | 12
  W24, Item 6, neutral, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 6, neutral, n=20;23 | 3 | 5
  W24, Item 6, like, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 6, like, n=20;23 | 6 | 6
  W48, Item 6, dislike, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 6, dislike, n=15;22 | 9 | 10
  W48, Item 6, neutral, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 6, neutral, n=15;22 | 1 | 6
  W48, Item 6, like, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 6, like, n=15;22 | 5 | 6
  W2, Item 7, no problem taking FPV, n=23;27 | 7 | 6
  W2, Item 7, few problems taking FPV, n=23;27 | 9 | 9
  W2, Item 7, problem taking most of time, n=23;27 | 5 | 10
  W2, Item 7, impossible to take, n=23;27 | 2 | 2
  W24, Item 7, no problem taking FPV, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 7, no problem taking FPV, n=20;23 | 13 | 10
  W24, Item 7, few problems taking FPV, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 7, few problems taking FPV, n=20;23 | 3 | 5
  W24, Item 7, problem taking most of time, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 7, problem taking most of time, n=20;23 | 4 | 8
  W24, Item 7, impossible to take, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 7, impossible to take, n=20;23 | 0 | 0
  W48, Item 7, no problem taking FPV, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 7, no problem taking FPV, n=15;22 | 8 | 10
  W48, Item 7, few problems taking FPV, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 7, few problems taking FPV, n=15;22 | 4 | 8
  W48, Item 7, problem taking most of time, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 7, problem taking most of time, n=15;22 | 2 | 2
  W48, Item 7, impossible to take, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 7, impossible to take, n=15;22 | 1 | 2
  W2, Item 8, swallows with no problem, n=23;27 | 9 | 10
  W2, Item 8, swallows with struggle, n=23;27 | 11 | 10
  W2, Item 8, spits out suspension, n=23;27 | 0 | 5
  W2, Item 8, vomits the suspension, n=23;27 | 3 | 2
  W24, Item 8, swallows with no problem, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 8, swallows with no problem, n=20;23 | 10 | 12
  W24, Item 8, swallows with struggle, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 8, swallows with struggle, n=20;23 | 7 | 9
  W24, Item 8, spits out suspension, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 8, spits out suspension, n=20;23 | 3 | 2
  W24, Item 8, vomits the suspension, n=20;23: number analyzed (Participants) | 20 | 23
  W24, Item 8, vomits the suspension, n=20;23 | 0 | 0
  W48, Item 8, swallows with no problem, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 8, swallows with no problem, n=15;22 | 11 | 12
  W48, Item 8, swallows with struggle, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 8, swallows with struggle, n=15;22 | 3 | 8
  W48, Item 8, spits out suspension, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 8, spits out suspension, n=15;22 | 1 | 1
  W48, Item 8, vomits the suspension, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 8, vomits the suspension, n=15;22 | 0 | 1
  W2, I9, take more willingly than other med., n=23;27 | 3 | 3
  W2, Item 9, about the same, n=23;27 | 13 | 15
  W2, I9, not as willing to take as other med., n=23;27 | 7 | 9
  W24, I9, take more willingly than other med., n=20;22: number analyzed (Participants) | 20 | 22
  W24, I9, take more willingly than other med., n=20;22 | 3 | 1
  W24, Item 9, about the same, n=20;22: number analyzed (Participants) | 20 | 22
  W24, Item 9, about the same, n=20;22 | 11 | 20
  W24, I9, not as willing to take as other med, n=20;22: number analyzed (Participants) | 20 | 22
  W24, I9, not as willing to take as other med, n=20;22 | 6 | 1
  W48, I9, take more willingly than other med., n=15;22: number analyzed (Participants) | 15 | 22
  W48, I9, take more willingly than other med., n=15;22 | 5 | 6
  W48, Item 9, about the same, n=15;22: number analyzed (Participants) | 15 | 22
  W48, Item 9, about the same, n=15;22 | 10 | 14
  W48, I9, not as willing to take as other med, n=15;22: number analyzed (Participants) | 15 | 22
  W48, I9, not as willing to take as other med, n=15;22 | 0 | 2
  Week 2, Item 10, dislike, n=23;27 | 11 | 9
  Week 2, Item 10, neutral, n=23;27 | 5 | 9
  Week 2, Item 10, like, n=23;27 | 7 | 9
  Week 24, Item 10, dislike, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, Item 10, dislike, n=20;24 | 7 | 13
  Week 24, Item 10, neutral, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, Item 10, neutral, n=20;24 | 2 | 7
  Week 24, Item 10, like, n=20;24: number analyzed (Participants) | 20 | 24
  Week 24, Item 10, like, n=20;24 | 11 | 4
  Week 48, Item 10, dislike, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, Item 10, dislike, n=15;22 | 7 | 8
  Week 48, Item 10, neutral, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, Item 10, neutral, n=15;22 | 4 | 7
  Week 48, Item 10, like, n=15;22: number analyzed (Participants) | 15 | 22
  Week 48, Item 10, like, n=15;22 | 4 | 7

42. Secondary Outcome: Correlation Between Steady-state Plasma APV PK Parameters to Changes in Plasma HIV-1 RNA Concentrations, CD4+ Percentages, and/or the Occurrence of Adverse Events
Description: No formal analysis has been performed or is planned to correlate plasma APV PK with efficacy and safety outcomes.
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Plasma FPV AUC (0-τ)
Description: The majority of the FPV data were below the quantification limit. Therefore, plasma FPV PK parameters were not estimated.
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Plasma FPV Cmax and Cτ
Description: as for outcome 43
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Plasma FPV CL/F Expressed in mL/Min/kg
Description: as for outcome 43
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: Plasma FPV CL/F Expressed in mL/Min
Description: as for outcome 43
Time Frame: Week 48
Population: PK Population
Arm/Group | FPV/RTV BID: 4 Weeks to <6 Months | FPV/RTV BID: 6 Months to <2 Years
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 684 weeks.
Description: All participants received FPV or FPV/RTV at any dose were included in the safety population.
Arm/Group | Cohort 2, Arm A - 4 Weeks to <6 Months | Cohort 1, Arm A - 6 Months to <2 Years
All-Cause Mortality (participants affected / at risk) | 1/29 | 2/30
Serious Adverse Events (participants affected / at risk) | 13/29 | 12/30
Other Adverse Events (participants affected / at risk) | 24/29 | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2, Arm A - 4 Weeks to <6 Months (N=29) | Cohort 1, Arm A - 6 Months to <2 Years (N=30)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal symptom (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Greenstick fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Herbal toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Kwashiorkor (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2, Arm A - 4 Weeks to <6 Months (N=29) | Cohort 1, Arm A - 6 Months to <2 Years (N=30)
Otorrhoea (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dental caries (Gastrointestinal disorders) | 6 (6) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 19 (19) | 15 (15)
Vomiting (Gastrointestinal disorders) | 8 (8) | 8 (8)
Pyrexia (General disorders) | 0 (0) | 5 (5)
Abdominal infection (Infections and infestations) | 3 (3) | 0 (0)
Acarodermatitis (Infections and infestations) | 4 (4) | 3 (3)
Bronchiolitis (Infections and infestations) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2)
Conjunctivitis (Infections and infestations) | 8 (8) | 3 (3)
Folliculitis (Infections and infestations) | 2 (2) | 1 (1)
Fungal skin infection (Infections and infestations) | 4 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 14 (14) | 7 (7)
Helminthic infection (Infections and infestations) | 5 (5) | 2 (2)
Impetigo (Infections and infestations) | 8 (8) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (7) | 10 (10)
Oral candidiasis (Infections and infestations) | 2 (2) | 2 (2)
Oral herpes (Infections and infestations) | 2 (2) | 5 (5)
Otitis media (Infections and infestations) | 7 (7) | 11 (11)
Otitis media acute (Infections and infestations) | 4 (4) | 4 (4)
Pharyngitis (Infections and infestations) | 8 (8) | 13 (13)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 2 (2)
Rhinitis (Infections and infestations) | 9 (9) | 11 (11)
Skin infection (Infections and infestations) | 3 (3) | 0 (0)
Tinea capitis (Infections and infestations) | 7 (7) | 2 (2)
Tinea infection (Infections and infestations) | 4 (4) | 0 (0)
Tonsillitis (Infections and infestations) | 9 (9) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 12 (12)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Blood cholesterol (Investigations) | 4 (4) | 2 (2)
Blood cholesterol increased (Investigations) | 7 (7) | 6 (6)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2)
Blood triglycerides increased (Investigations) | 4 (4) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Herpes simplex (Infections and infestations) | 2 (2) | 0 (0)
Measles (Infections and infestations) | 2 (2) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 2 (2) | 0 (0)
Mumps (Infections and infestations) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 1 (1)
Viral rash (Infections and infestations) | 0 (0) | 2 (3)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Candida nappy rash (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Erythema infectiosum (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0)
Tinea faciei (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood sodium increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Underweight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Developmental delay (General disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Eye allergy (Eye disorders) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ichthyosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immunisation reaction (Immune system disorders) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Educational problem (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT00071760/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT00071760/SAP_001.pdf